CLINICAL TRIAL: NCT02355639
Title: A Single-Centre, Explorative, Randomised, Investigator-Blinded, Negative-Controlled, Phase I Clinical Trial With Intra-Individual Comparison of Treatments to Assess Steroid Induced Skin Atrophy on Healthy Skin
Brief Title: A Single-Centre Clinical Trial to Assess Steroid Induced Skin Atrophy on Healthy Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EXP-1090
Record Dates: First submitted 2015-01-27; First posted 2015-02-04 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2017-05

CONDITIONS: Skin and Connective Tissue Diseases
MeSH Terms: conditions — Skin and Connective Tissue Diseases | interventions — Clobetasol; Ointments; betamethasone-17,21-dipropionate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clobetasol propionate 0.05 % ointment (Experimental): Active drug
  Interventions: Drug: Clobetasol propionate 0.05 % ointment
- Betamethasone dipropionate 0.064 % ointment (Experimental): Active drug
  Interventions: Drug: Betamethasone dipropionate 0.064 % ointment
- Petrolatum ointment (Placebo Comparator): Placebo drug
  Interventions: Drug: Petrolatum ointment

INTERVENTIONS:
Drug: Clobetasol propionate 0.05 % ointment
  Arms: Clobetasol propionate 0.05 % ointment
Drug: Betamethasone dipropionate 0.064 % ointment
  Arms: Betamethasone dipropionate 0.064 % ointment
Drug: Petrolatum ointment
  Arms: Petrolatum ointment

SUMMARY:
The purpose of this study is to assess steroid induced skin atrophy by sonography.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, 25 to 40 years old inclusive.
2. Healthy skin on volar arms with a hairless area sufficient for measurements

Exclusion Criteria:

1. Clinical skin atrophy, telangiectasia or striae on volar arms.
2. Presence of any skin condition or colouration that would interfere with test sites or the response or assessment.
3. Fitzpatrick skin type IV - VI.
4. History or current evidence of infection, eczema or other relevant skin disease.

Ages: 25 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in skin thickness from baseline to end of treatment | 4 weeks

SECONDARY OUTCOMES:
Relation of clinical features (skin transparency and telangiectasia) to the steroid induced skin atrophy after end of treatment | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitaetsmedizin Berlin, Department of Dermatology and Allergy, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en